CLINICAL TRIAL: NCT07235462
Title: ACO-REAL - A Non-interventional Study Providing Insights Into the Use of Acoramidis in Patients With ATTR Amyloidosis With Cardiomyopathy (ATTR-CM) in Routine Clinical Practice
Brief Title: A Study to Learn About the Use of Acoramidis in Patients With a Heart Condition Called Transthyretin Amyloid Cardiomyopathy (ATTR-CM) in a Real-world Setting
Acronym: ACO-REAL
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 23023
Record Dates: First submitted 2025-10-06; First posted 2025-11-19 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Transthyretin Amyloid Cardiomyopathy (ATTR-CM)
Keywords: Transthyretin Amyloidosis; Cardiomyopathy; Heart Failure; Wild-type Amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Cardiomyopathies; Heart Failure | interventions — attruby

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acoramidis Arm: Patients with Transthyretin Amyloid Cardiomyopathy (ATTR-CM) initiating treatment with acoramidis in routine clinical practice.
  Interventions: Drug: Acoramidis (356 mg film-coated tablets)

INTERVENTIONS:
Drug: Acoramidis (356 mg film-coated tablets) — Follow clinical practice/administration.
  Other Names: BEYONTTRA

SUMMARY:
Transthyretin Amyloid Cardiomyopathy (ATTR-CM) is a serious and life-threatening condition where a protein called transthyretin (TTR) misfolds and builds up as amyloid fibrils in the heart muscle. This buildup causes the heart to become stiff, leading to restrictive cardiomyopathy and progressive heart failure. There are two forms of ATTR-CM: a hereditary or 'variant' form (vATTR-CM) caused by a gene mutation, and a 'wild-type' form (wtATTR-CM) which is associated with aging. Because its symptoms can be similar to other heart conditions, ATTR-CM is often diagnosed late. However, recent advances in medical imaging are helping doctors to identify the disease earlier. Acoramidis is a new medication designed to treat ATTR-CM. It works by stabilizing the TTR protein, preventing it from misfolding and forming the harmful amyloid deposits. Acoramidis has been shown to be effective and safe in a major clinical trial (the ATTRibute-CM study), which led to its approval for use in both the United States and Europe. While clinical trials provide valuable information, data on how a new medicine performs in everyday clinical practice is also very important. This type of information is called real-world evidence. Currently, there is limited real-world information about the use of acoramidis. This study, called ACO-REAL, is an observational study, which means researchers will observe patients who are receiving acoramidis as part of their normal clinical care, without introducing any experimental interventions. The study will take place in approximately 20 European countries and aims to enroll up to 2,000 adults who have been diagnosed with either wild-type or variant ATTR-CM and are starting treatment with acoramidis. This includes patients who have not been treated for ATTR-CM before, as well as those who have been treated with other therapies. The main goals of the study are to understand the characteristics of patients being treated with acoramidis and to document how the treatment is used in routine medical practice. The study will also collect information on the safety of acoramidis. Furthermore, researchers will assess how the treatment affects patients' heart function, their functional capacity (such as their ability to walk), their overall health status, and their quality of life. The study will also track how often patients need to use healthcare resources like hospitals or emergency rooms. This information will help to improve the understanding and management of ATTR-CM in a real-world setting, ultimately aiming to optimize care for patients with this progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* - Adults (≥18 years at the date of signing the informed consent form (ICF)).
* Diagnosis of either wild-type or variant ATTR-CM.
* Signed ICF.
* Decision to initiate treatment with acoramidis was made as per treating investigator's routine treatment practice before signature of ICF.
* Treatment start with acoramidis within 90 days after signing the ICF, with the possibility of starting acoramidis on the same day as signing the ICF.

Exclusion Criteria:

* Participation in an investigational trial with interventions outside of routine clinical practice, except for participation in potential sub-studies related to this observational study. Please note: In addition to this observational study, separate sub-studies may be conducted to collect additional data. Participation in these sub-studies is voluntary and will be governed by separate protocols and informed consent processes. The main observational study does not include interventional procedures beyond routine clinical practice.

  * Contra-indications according to the local SmPC of acoramidis.
  * Patients who are unable to provide consent, including those whose consent would need to be given by a legal representative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an established diagnosis of either wild-type or variant Transthyretin Amyloid Cardiomyopathy (ATTR-CM) who are eligible for treatment with acoramidis based on the clinical decision of the investigator, made independently of the study.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-03 (Estimated)

PRIMARY OUTCOMES:
Patient demographic characteristics: age | Baseline (Initial study visit)
  Demographic characteristics at the first documented regular visit in the study, referred to as the initial study visit.
Patient demographic characteristics: sex | Baseline (Initial study visit)
  Demographic characteristics at the first documented regular visit in the study, referred to as the initial study visit.
Patient demographic characteristics: race | Baseline (Initial study visit)
  Demographic characteristics at the first documented regular visit in the study, referred to as the initial study visit.
Patient demographic characteristics: height | Baseline (Initial study visit)
  Demographic characteristics at the first documented regular visit in the study, referred to as the initial study visit.
Patient demographic characteristics: weight | Baseline (Initial study visit)
  Demographic characteristics at the first documented regular visit in the study, referred to as the initial study visit.
Clinical Characteristics: Transthyretin Amyloid Cardiomyopathy (ATTR-CM) Type | Baseline up to 15 months
  ATTR-CM type: mixed phenotype (yes/no)
Clinical Characteristics: Transthyretin Amyloid Cardiomyopathy (ATTR-CM) Genetic status | Baseline up to 15 months
  ATTR-CM type: genetic status (mutation / wild type; if mutation: genotype and zygosity)
Clinical Characteristics: Transthyretin Amyloid Cardiomyopathy (ATTR-CM) Diagnosis | Baseline up to 15 months
  ATTR-CM diagnosis (year of diagnosis)
Clinical Characteristics: Transthyretin Amyloid Cardiomyopathy (ATTR-CM) Setting of Diagnosis | Baseline up to 15 months
  ATTR-CM setting of diagnosis: (endomyocardial biopsy
  / non-invasive / both, NYHA classification at diagnosis)
Clinical Characteristics: Transthyretin Amyloid Cardiomyopathy (ATTR-CM) Manifestations | Baseline up to 15 months
  ATTR-CM manifestations (type)
Clinical Characteristics: Transthyretin Amyloid Cardiomyopathy (ATTR-CM) -relevant comorbidities | Baseline up to 15 months
  ATTR-CM-relevant comorbidities (type)
Clinical Characteristics: Transthyretin Amyloid Cardiomyopathy (ATTR-CM) -relevant procedures | Baseline up to 15 months
  Prior and concomitant ATTR-CM-relevant procedures (type)
Treatment Patterns with Acoramidis: Transthyretin Amyloid Cardiomyopathy (ATTR-CM) -related medications | Baseline (assessment within the past 12 months prior to initiation)
  Previously administered ATTR-CM-related medications within the past 12 months before initial visit (name)
Treatment Patterns with Acoramidis: Transthyretin Amyloid Cardiomyopathy (ATTR-CM) concomitant medications | Baseline up to 15 months
  Concomitant medications administered alongside acoramidis (name)
Treatment Patterns with Acoramidis: Initiation | Baseline up to 15 months
  Acoramidis initiation (date)
Treatment Patterns with Acoramidis: Initiation after a different therapy | Baseline up to 15 months
  Acoramidis initiation (if patient is switching from a different therapy: reason for switch)
Treatment Patterns with Acoramidis: discontinuation | Baseline up to 15 months
  Acoramidis discontinuation (reason)
Treatment Patterns with Acoramidis: interruption | Baseline up to 15 months
  Acoramidis interruption (reason)
Treatment Patterns with Acoramidis: prescription / refills | Baseline up to 15 months
  Acoramidis prescriptions/refills since the last visit or telephone contact (duration of time from initiation to discontinuation of therapy)

SECONDARY OUTCOMES:
Incidence of Adverse Events | From acoramidis initiation up to end of observation (approximately 12-15 months).
  Adverse events (AEs) documentation
Incidence of Serious Adverse Events | From acoramidis initiation up to end of observation (approximately 12-15 months).
  Serious Adverse events (SAEs) documentation

CONTACTS AND LOCATIONS:
Locations (1):
- Universitaetsklinik Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.